CLINICAL TRIAL: NCT00252200
Title: Low Dose Continuous Infusion of BNP (Nesiritide) in the Prevention of Renal Insufficiency Post Cardiopulmonary Bypass Cardiac Surgery.
Brief Title: BNP (Nesiritide) vs. Placebo to Protect Kidney Function in Patients Undergoing Heart Bypass Surgery.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Horng H. Chen, Mayo Clinic Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 621-03
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Acute Kidney Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Neseritide — Dose of Nesiritide infusion will be 0.005 ug/Kg/min
  Other Names: BNP, Nesiritide

SUMMARY:
Use of BNP (nesiritide) vs placebo to help protect kidney function in patients undergoing heart bypass surgery.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study of low dose nesiritide to prevent renal insufficiency after cardiopulmonary bypass surgery. Patients included are those with greater than mild renal insufficiency preoperatively as defined by having a creatinine clearance of less than 50 mL/minute determined by the Cockroft-Gault formula. The infusion of nesiritide (BNP) 0.005 mcg/Kg/minute or placebo begins 1 hour before surgery and runs for 24 hours started after the induction of anesthesia prior to cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old, undergoing cardiac surgery requiring cardiopulmonary bypass with baseline creatinine clearance < 50 ml/min and who are not dialysis dependent.

Exclusion criteria:

* Cardiogenic shock or hypotension with systolic BP < 90 mmHg.
* Patients with acute or chronic aortic dissection.
* Patients who are enrolled in other studies that have an effect the renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Creatinine Clearance at 72 hours determined by the Cockroft-Gault formula | 72 hours post op

SECONDARY OUTCOMES:
Number of patients requiring dialysis during the hospitalization | before hospital discharge
Plasma aldosterone levels at 12 hours and 24 hours | 12 hours and 24 hours postoperatively
Total time on ventilator, ICU length of stay, total length of stay in hospital | total length of hospital stay
pre and postoperative diuretic dose used | pre operative and postoperate
Need or absence of need for inotropic support in the 72 hour perioperative period | 72 hours perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States